CLINICAL TRIAL: NCT05894304
Title: The Effects of Scapular Muscles Training Using a Suspension System in Patients With Non Spacific Chronic Neck Pain and Scapular Dyskinesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Gamal Khattab, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004031
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Scapular Dyskinesis
Keywords: Scapular diskinesia; Non spacific chronic neck pain; Suspension system

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Excercise therapy group (Active Comparator): The group that recived scapular muscle training exercises
  Interventions: Other: Scapular training exercises
- Suspension group (Experimental): The group that recived scapular muscle training using suspension system
  Interventions: Device: Suspension system

INTERVENTIONS:
Device: Suspension system — suspended from the handles of the straps by either their hands or feet while the non-suspended pair of extremities are in contact with the ground leading to muscle activation due to unstable base of support
  Other Names: Sling therapy
  Arms: Suspension group
Other: Scapular training exercises — Scapular muscle strength by resistance
  Arms: Excercise therapy group

SUMMARY:
The study aimed to investigate the effect of scapular muscle training using a suspension system in patients with non spacific chronic neck pain with scapular diskinesia

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 20-35 years.
* Patients with non spacific pain(pain > 3 month).
* pain must have been present for at least the previous 12 weeks.
* Patients with non spacific chronic neck pain with scapular dyskinesia.
* Patient BMI<30.

Exclusion Criteria:

* History of previous neck surgery.
* Recent or old fractures.
* Cognitive impairment and inability to understand the scale.
* Systematic inflammatory disease e.g., rheumatoid arthritis and ankylosing Spondylitis.
* Neck pain with radiculopathy or neuropathy.
* Scapular dyskinesia due to other pathology such as shoulder impingement

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 1week
  Pain intensity is measured by neumeric pain rating scale the lowest value is 0 means no pain and the highest value is 10 means the worst pain
Function | 1 week
  Function is measured by neck disability index the total score is 50 as the score is higher the disability is higher
Scapular muscle strength | 1week
  Scapular muscle strength is measured by hand held dynanometer
Scapular position | 1week
  Scapular position is measured by lateral scapular slide test

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes